CLINICAL TRIAL: NCT03247621
Title: External Eating: An Investigation of Social Media and Environmental Factors Influencing Eating Behaviours
Brief Title: Exploring the Effects of Social Media Use and Environmental Factors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yale-NUS College (Other)
Collaborators: Raffles Institution (Other)
Responsible Party: Principal Investigator, Jean Liu, Assistant Professor, Yale-NUS College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A-15-170
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Whatsapp, Article, No Phone
Keywords: external eating, technology
MeSH Terms: interventions — Household Articles

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whatsapp (Experimental): Participants will engage in Whatsapp chats on their smartphones during the taste test
  Interventions: Behavioral: Whatsapp
- Article (Placebo Comparator): Participants will read a neutral article on their smartphones during the taste test
  Interventions: Behavioral: Article
- No Phone (Active Comparator): Participants will not use their phones during the taste test
  Interventions: Behavioral: No Phone

INTERVENTIONS:
Behavioral: Whatsapp
  Arms: Whatsapp
Behavioral: Article
  Arms: Article
Behavioral: No Phone
  Arms: No Phone

SUMMARY:
In this protocol, the investigators propose a randomised controlled trail to explore the effects of environmental factors and the use of technology on eating behaviours. The investigators have planned two studies to investigate these effects, one on high school students from Raffles Institution, and the other on the university population in the National University of Singapore.

DETAILED DESCRIPTION:
Participants will be told a cover story that the study explores technological distraction on taste, and asked to complete a taste-evaluation taste of common snacks. One group (intervention group) will be asked to use their personal smartphones to engage in their pre-existing Whatsapp chats while doing the taste test. For the two control conditions, one group will be tasked with reading a neutral article on their personal smartphones while they complete the taste test, while the other group will be asked to complete the taste test without any use of smartphones.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight: Body mass index of 18 to 25
* Have at least occasional breakfast meals (≥ 3 times a week of self-reported consumption of a breakfast meal)

Exclusion Criteria:

* Symptoms / history of any medical or psychiatric conditions
* Allergies to food products
* History of eating disorders
* Excessive exercise (≥ 5 times a week of self-reported exercise)
* Currently on a special diet or deliberating restricting caloric intake
* Currently on a weight loss program
* Smoking or substance abuse

Ages: 13 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Amount of food consumed | 20 minutes
  Number of grams of cereal eaten

SECONDARY OUTCOMES:
Hunger ratings | 10 minutes
  Self-reported hunger ratings before and after the taste test
Taste ratings | 20 minutes
  Self-report on how much they enjoyed the two food products during the taste test

CONTACTS AND LOCATIONS:
Locations (1):
- Yale-NUS College, Singapore, Singapore